CLINICAL TRIAL: NCT05095766
Title: Differentiation Between Radionecrosis and Tumor Recurrence for Post-stereotactic Radiosurgery Follow-up by Pharmacokinetic Analyses in Perfusion MRI and Positron Emission Tomography
Brief Title: Comparaison Between MRI Alone or Combined With Positron Emission Tomography for Brain Metastasis Diagnosis
Acronym: ITIRR
Status: Completed | Type: Observational
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-1488
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Brain Metastases, Adult
Keywords: Magnetic resonance imaging; Radiofrequency; Radionecrosis; Tumor recurrence; Post-stereotactic surgery; Positron emission tomography; CT scan; 18F-fluoroethyl-tyrosine; Perfusion MRI
MeSH Terms: conditions — Brain Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During gamma scalpel treatment of brain tumors and metastases, a follow-up magnetic resonance imaging (MRI) scan is performed. The radiologist who reviews the MRI assesses whether there is an increase in signal at the tumor site. This increase potentially indicates that the treatment was not effective. However, in 25% of cases (one in four people), this signal enhancement is not due to ineffective treatment, but to inflammation (swelling/damage) and tissue death around the tumor. This is why when an increase in signal is detected, additional follow-up is essential. The standard additional follow-up has an accuracy of about 83%.

This is an observational study on patients with brain metastatis comparing MRI alone or combined to PET-FET to improve accuracy of diagnosis of metastasis recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age;
* Having undergone gamma knife radiosurgery for brain metastasis;
* Presenting for a first MRI follow-up (Cohort C1);
* Presence of one or more brain metastases with increased enhancement on follow-up MRI (Cohort C2.1 and C2.2); A participant recruited for Cohort C1 could be recruited for follow-up in Cohort C2.1 or C2.2 if the MRI result is ambiguous.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Other condition that may influence the imaging result;
* Renal impairment (<30 mL/min/1.73 m2). This threshold is consistent with recent RAC recommendations; Note: For participants with intermediate renal clearance (30-60 mL/min/1.73 m2), the total gadobutrol dose injected is set at the manufacturer's recommended clinical dose. For patients with renal clearance greater than 60 mL/min/1.73 m2, a dose of 1.5x the normal dose is used. These dose values have been approved by Dr. Chénard and are consistent with the RAC recommendations.
* Inability to maintain supine position for the required duration (variable, depending on the sequence);
* Patients who have previously received full brain irradiation;
* Patients who are claustrophobic and cannot tolerate insertion into the MRI scanner;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with brain metastases undergoing MRI
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Comparison of novel MRI method with current MRI exam method | Following MRI exam
  In the context of differentiating radionecrosis and recurrence of metastasis: Is our new method better than the actual standard of care in Sherbrooke?
Comparison of DCE-MRI method with FET PET | Following MRI exam
  In the context of differentiating radionecrosis and recurrence of metastasis: is one better than the other? And Can DCE-MRI and FET PET be combined to differentiate between recurrence/radionecrosis?

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No